CLINICAL TRIAL: NCT07323563
Title: A Randomized, Crossover, Confinement Study to Assess Nicotine Uptake From Electronic Nicotine Delivery System Products
Brief Title: A Study to Assess Nicotine Uptake From Electronic Nicotine Delivery Systems
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CSD252102
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Smoking; Smoking Behaviors; Tobacco Use; Tobacco Smoking
MeSH Terms: conditions — Smoking; Tobacco Use; Tobacco Smoking | interventions — HTR3D protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Product usage order AHBGCFDE (Experimental): Subjects will use each of the 8 products during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product H
- Product usage order BACHDGEF (Experimental): Subjects will use each of the 8 products during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product H
- Product usage order CBDAEHFG (Experimental): Subjects will use each of the 8 products during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product H
- Product usage order DCEBFAGH (Experimental): Subjects will use each of the 8 products during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product H
- Product usage order EDFCGBHA (Experimental): Subjects will use each of the 8 products during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product H
- Product usage order FEGDHCAB (Experimental): Subjects will use each of the 8 products during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product H
- Product usage order GFHEADBC (Experimental): Subjects will use each of the 8 products during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product H
- Product usage order HGAFBECD (Experimental): Subjects will use each of the 8 products during an evaluation period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F; Other: Product G; Other: Product H

INTERVENTIONS:
Other: Product A — Menthol Flavor, 5%
  Other Names: P2611222
Other: Product B — Mint Flavor, 5%
  Other Names: P2615422
Other: Product C — Tobacco Flavor, 5%
  Other Names: P2615222
Other: Product D — Fruit Flavor, 5%
  Other Names: P2615022
Other: Product E — Fruit Flavor, 5%
  Other Names: P2615522
Other: Product F — Fruit Flavor, 5%
  Other Names: P2612222
Other: Product G — Fruit Flavor, 5%
  Other Names: P2615622
Other: Product H — Fruit Flavor, 5%
  Other Names: P2615122

SUMMARY:
This will be an open-label, randomized, single-site, 8-way crossover study designed to evaluate plasma nicotine pharmacokinetic (PK) parameters and overall product liking (OPL) following an ad libitum use of Electronic Nicotine Delivery System (ENDS) investigational products (IPs) in a confinement setting by generally healthy adult combustible cigarette smokers and smokers who also use ENDS products.

DETAILED DESCRIPTION:
This study is designed to evaluate plasma nicotine PK parameters and OPL following use of ENDS IPs in generally healthy adult menthol or nonmenthol cigarette smokers and smokers who also use ENDS. A summary of study activities is provided below:

Potential participants will undergo a pre-screening interview followed by a Screening Visit to assess their eligibility. The screening assessments will occur within 28 days prior to enrollment, randomization, and study confinement.

Following the Screening Visit, eligible participants will be scheduled for a Checkin and Randomization visit. At this visit, participants' continued eligibility will be confirmed before participants are randomized to a product use sequence and begin a confinement period of 9 nights and 10 days.

Beginning on Study Day 1, participants will start a ENDS IP familiarization period. During this period, participants will be required to use 3 ENDS IPs (Product A , Product B, and Product D) at least once for approximately 5 minutes, following which they will be permitted ad libitum smoking of their usual-brand (UB) cigarettes. Participants who also use other tobacco- and/or nicotine-containing products such as ENDS, smokeless tobacco, or modern oral nicotine products in addition to their UB cigarettes will not have access to those products during the study.

Starting on Day 3, participants will participate in 8 separate test sessions (1 test session per day) to assess nicotine PK and OPL, with 1 session conducted for each ENDS IP. Beginning on Day 2 and each day prior to a subsequent test session, participants will undergo a product acclimation period during which they will use their assigned ENDS IP at least 4 times for approximately 5 minutes each use, in preparation for the following day's test session. Following this acclimation use, participants will be permitted ad libitum smoking of their UB cigarettes. The site will capture information on product usage during the product familiarization and acclimation periods.

At the end of the product acclimation period and ad libitum use of the participant's UB cigarette, participants will abstain from use of all tobacco and nicotine-containing products for a minimum of 12 hours prior to each test session occurring on the following day. In addition, participants will be required to abstain from any caffeine-containing products for 4 hours prior to the start of each test session through the end of the test session.

From Day 3 through Day 10, each participant will complete 8 test sessions, 1 per day, each lasting approximately 4 hours and evaluating 1 ENDS IP per session. During each test session, blood samples will be collected for nicotine PK assessments and participants will complete the OPL questionnaires.

Each session will begin with an approximately 5-minute ad libitum use of a single ENDS IP. The order of the ENDS IPs used during these 8 test sessions will be determined by a randomized 8-sequence presentation schedule generated using a Williams Design. Each test session will be preceded by a 12hour abstention from all tobacco- and nicotine-containing products.

Participants' use of the ENDS IP will be self-defined during the 5minute ad libitum IP use session; specific parameters around puff duration, volume, inter-puff interval, and quantity will not be prescribed.

ENDS IP cartridges will be weighed within 4 hours before and after the test session on Days 3 to 10.

Safety will be monitored throughout the study by the Principal Investigator (PI) (or qualified designee) by assessing adverse events (AEs), vital sign measurements, physical examinations (including an oral examination), and clinical laboratory tests. The Medical Monitor will be available for consultation during the duration of the study and for any follow-ups after study discharge

ELIGIBILITY:
Inclusion Criteria:

* Able to read, understand, and willing to sign an informed consent form (ICF) and complete questionnaires written in English.
* Generally healthy male or female, 21 to 60 years of age, inclusive, at the time of consent.
* Expired breath carbon monoxide (ECO) level is ≥ 10 ppm and ≤ 100 ppm at Screening.
* Positive urine cotinine test at Screening.
* Smokes combustible, filtered, menthol or non-menthol cigarettes, 83 mm to 100 mm in length.
* Agrees to smoke same UB cigarette throughout the study period. UB cigarette is defined as the cigarette brand style currently smoked most frequently by the participant.
* Participants must meet one (a or b) of the following tobacco use conditions:

  1. Smokes at least 10 cigarettes per day (on average) and inhales the smoke, for at least 6 months prior to Screening. Brief periods of abstinence due to illness, quit attempt (more than 30 days prior to Screening), or clinical study participation (more than 30 days prior to Screening) will be allowed at the discretion of the Principal Investigator (PI).
  2. Dual user of cigarettes and ENDS who self-reports:

  i. Smoking at least 10 cigarettes per day (on average) and inhales the smoke, for at least 6 months prior to Screening. Brief periods of abstinence more than 30 days prior to Screening due to illness, quit attempt, or clinical study participation will be allowed at the discretion of the PI and ii. Using a nicotine-containing ENDS (cartridge or tank system). NOTE: Cigarette smokers or ENDS users who also use other tobacco- or nicotine-containing products (e.g., smokeless tobacco and modern oral nicotine products) on no more than 1 day per week will not be excluded from study participation.
* Response at Screening to the Fagerström Test for Nicotine Dependence (FTND) Question 1 ("How soon after you wake up do you smoke your first cigarette?") is either "Within 5 minutes" or "6-30 minutes."
* Willing to use only UB cigarette and assigned test ENDS IPs during the study period.
* Willing to abstain from tobacco and nicotine use for at least 12 hours prior to each test session.
* Females must be willing to use a form of contraception acceptable to an Investigator, including abstinence from heterosexual intercourse, from the time of signing informed consent until EOS. Examples of acceptable means of birth control include, but are not limited to:

  1. Surgical sterilization (hysterectomy, bilateral tubal ligation/occlusion, bilateral oophorectomy, bilateral salpingectomy);
  2. Physical barrier method (e.g., condom, diaphragm/sponge/cervical cap) with spermicide;
  3. Non-hormone-releasing intrauterine devices (IUDs) or hormone-releasing IUDs (e.g., Mirena or Kyleena);
  4. Vasectomized partner;
  5. Post-menopausal and not on hormone replacement therapy; or
  6. Sexual abstinence, defined as refraining from intercourse, when this is in line with the preferred and usual lifestyle of the participant.
* Males must use an acceptable method of birth control from Day 1 Check-in until EOS, unless they have had a vasectomy or are abstinent from heterosexual intercourse, or their female partner is not able to bear children.
* Agrees to in-clinic confinement of 10 days and 9 nights.

Exclusion Criteria:

* Presence of clinically significant uncontrolled cardiovascular, pulmonary, renal, hepatic, endocrine, gastrointestinal, psychiatric, hematological, neurological disease, or any other concurrent disease or medical condition that, in the opinion of the PI, makes the study participant unsuitable to participate in this clinical study.
* History, presence of, or clinical laboratory test results indicating diabetes.
* Systolic blood pressure of > 160 mmHg or a diastolic blood pressure of > 95 mmHg, measured after being seated for 5 minutes at Screening and at Check-in Day 1.
* Weight of ≤ 110 pounds (≤ 50.0 kg) and body mass index of > 40.0 kg/m2 at Screening.
* Hemoglobin level is < 12.5 for females or < 13.0 for males g/dL at Screening.
* Scheduled treatment for asthma currently or within the past consecutive 12 months prior to the Screening Visit. As-needed treatment, such as inhalers, may be included at the PI's discretion.
* Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
* Any history of cancer, except for primary cancers of skin such as localized basal cell/squamous cell carcinoma that has been surgically and/or cryogenically removed.
* Must not be a current regular user (i.e., > 5 times per month) of any tobacco- or nicotinecontaining products other than cigarettes or ENDS within the last 6 months prior to Screening.
* Use of any medication or substance that aids in smoking cessation, including but not limited to any NRT (e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), glucagon-like peptide-1 (GLP-1) agonists (e.g., Wegovy®, Mounjaro®, Ozempic®), or lobelia extract within ≤ 30 days prior to the signing of informed consent.
* History or presence of bleeding or clotting disorders.
* Use of daily aspirin (≥ 325 mg) or other daily anticoagulants.
* Whole blood donation within 8 weeks (≤ 56 days) prior to the signing of informed consent and between Screening and Check-in Day 1.

NOTE: Participants will be advised against scheduling a whole blood donation for at least 7 days following study completion.

• Plasma donation within ≤ 7 days prior to the signing of informed consent and between Screening and Check-in Day 1.

NOTE: Participants will be advised against scheduling a plasma donation for at least 7 days following study completion.

* Participation in another clinical trial within ≤ 30 days prior to the signing of informed consent. The 30-day window for each participant will be derived from the date of the last study event in the previous study to the time of signing the ICF in the current study.
* Females who have a positive pregnancy test at Screening or Check-in on Day 1, are pregnant, breastfeeding, or intend to become pregnant during the course of the study.
* Individuals ≥ 35 years of age currently using systemic, estrogen-containing contraception or hormone replacement therapy.
* Has positive urine drug screen or alcohol test (urine or breath) at Screening or at Checkin to the Assessment Phase (Day 1), with the exception of positive results for tetrahydrocannabinol (THC). If positive for THC at Check-in (Day 1), a cannabis intoxication evaluation will be performed, and inclusion will be at the discretion of an Investigator.
* Postpones a decision to quit using tobacco- or nicotine-containing products in order to participate in this study or a previous quit attempt within ≤ 30 days prior to the signing of the ICF.
* Has a significant history of alcoholism or drug abuse within 24 months prior to Screening, as determined by the PI, or has a positive alcohol test at Screening or Checkin on Day 1.
* Employed by a tobacco or nicotine company, the study site, or handles tobacco- or nicotine-containing products as part of their job.
* Individuals or their family members who have ongoing litigation with tobacco company(ies).
* Determined by the PI to be inappropriate for this study.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
AUC nic 0-240 | 0 to 240 minutes
  Baseline-adjusted area under the plasma nicotine concentration-versus-time curve from time zero to 240 minutes after the start of IP use
Cmax | 240 minutes
  Maximum baseline-adjusted plasma concentration of nicotine

CONTACTS AND LOCATIONS:
Overall Officials: Milly Kanobe, Study Director — Reynolds American

IPD SHARING:
Plan to Share IPD: No